CLINICAL TRIAL: NCT01983384
Title: A Randomised Controlled Trial to Reduce Postoperative Delirium Through Reduction in Intraoperative EEG Suppression in Older Surgical Patients Undergoing Major Noncardiac Surgery
Brief Title: Anesthetic Depth and Postoperative Delirium Trial - 2
Acronym: ADAPT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANESDEPTH
Record Dates: First submitted 2013-10-29; First posted 2013-11-14 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Delirium; Cognitive Disorders
Keywords: Delirium; Cognition; Surgery; Anesthesia; Aging; Electroencephalography
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to receive processed EEG-guided anesthesia or standard anesthetic care. Patients in both groups will be monitored with processed EEG, however those in the standard care group will have the anesthesiologist blinded to the machine. Patients in the interventional group receive processed EEG-guided anesthetic maintenance.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are assigned to study arm by random number generator. Anesthesiologists are informed which study arm the patient is assigned before the day of surgery. Patients are not informed of study arm assignment. Research staff assessing for postoperative delirium are not informed of patient study arm assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Anesthetic Depth: standard care (Placebo Comparator): A cohort of older patients undergoing major non-cardiac surgery will be randomized to receive routine anesthetic management not guided by the processed electroencephalogram
  Interventions: Other: Processed EEG-guided anesthetic depth
- Anesthetic Depth: interventional (Experimental): A cohort of older patients undergoing major non-cardiac surgery will be randomized to receive anesthetic management guided by the processed electroencephalogram (processed EEG-guided anesthetic depth)
  Interventions: Other: Processed EEG-guided anesthetic depth

INTERVENTIONS:
Other: Processed EEG-guided anesthetic depth — Investigators will undertake a randomized control trial in a cohort of older patients undergoing major non-cardiac surgery to receive either a control vs. an intervention of anesthesia as determined by a processed electroencephalogram

SUMMARY:
Recent limited evidence suggests that anesthetic depth may influence postoperative cognitive outcomes, however, the mechanism between this association is unclear.

DETAILED DESCRIPTION:
Recently, it has been proposed that use of a processed electroencephalogram (EEG) monitor during surgery may be associated with a lower rate of postoperative delirium. In fact, some suggest that older patients undergoing surgery should routinely be monitored with an anesthetic depth monitor to allow the titration of anesthetics or sedation medications to lighter levels to promote better postoperative cognitive outcomes. Recent studies, including preliminary results from our group, have demonstrated electroencephalogram (EEG) suppression to be an independent risk factor for postoperative delirium.

Prior studies that have focused on risk prediction have shown age and prior cognitive impairment to be the most consistent risk factors for postoperative delirium. However, as of yet, no clinical trial has identified a relationship whether use of processed EEG monitor resulted in a reduction of incident postoperative delirium through a reduction in EEG suppression, with proper consideration of patients' baseline cognitive status as a potential moderator. Additionally, use of anesthetic depth monitor to keep patients' anesthetic depth above a specified value has never been validated or proven to be feasible or safe.

Accordingly, the investigators plan an exploratory study to: 1) determine whether the use of processed EEG to keep anesthetic depth above a specified level, results in a reduction in EEG suppression when compared to standard anesthetic care, 2) to determine whether preoperative level of cognitive function moderates the effect of group assignment on EEG suppression, and 3) to determine the feasibility and safety of using processed EEG-guided to keep patients' anesthetic depth above a specified value. A secondary aim was to determine the effect size for the intervention to reduce postoperative delirium for subjects with and without preoperative cognitive impairment for a future trial.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older of age undergoing non-cardiac surgery, requiring hospital stay of 2 or more days.

Exclusion Criteria:

* patients who are not fluent in English or cannot provide informed consent
* patients who may not tolerate either light or deep anesthesia (history of heart failure, coronary artery disease, substance abuse)
* history of intraoperative recall or awareness during anesthesia
* pathologies of the brain which may affect EEG monitoring
* patients who are anticipated to have consecutive surgery within 3 days of first procedure
* patients who have had surgery with general anesthesia in the past 30 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 205 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative EEG Suppression | Patients will be monitored by processed EEG intraoperatively, for the duration of surgery
  Intraoperative EEG suppression will be measured by processed EEG monitor

SECONDARY OUTCOMES:
Preoperative level of cognitive function | Up to one week before surgery
  Level of cognitive function will be measured by Telephone Interview for Cognitive Status
Patient intraoperative awareness and recall | Intraoperative recall and awareness will be measured within 72 hours after end of surgery
  Intraoperative recall and awareness measured using modified Brice questionnaire (2 question survey - each answered with a yes or no, with additional checkboxes for applicable descriptions of events recalled [e.g. "Hearing voices," "Feeling pain," etc]) Patients answering yes to either question are classified as accidental awareness after general anesthesia (AAGA), which is regarded as an intraoperative adverse event.
Patient movement | During surgery
  Patient movement will be recorded from the anesthesia record
Intraoperative systolic and diastolic blood pressure | During surgery
  Intraoperative systolic and diastolic blood pressure will be continuously downloaded onto a computer for subsequent analysis. Increases or decreases above the preoperative baseline measurements will be measured and recorded from the medical record
Intraoperative heart rate | During surgery
  Intraoperative heart rate will be continuously downloaded onto a computer for subsequent analysis. Increases or decreases above the preoperative baseline measurements will be measured and recorded from the medical record
Anesthesiologists' adherence to assigned processed EEG index in the interventional group | Anesthesiologists complete self-report within 72 hours after end of surgery. This outcome measure is collected once for each patient through study completion, an average of 2 years.
  Anesthesiologists' assigned to patients randomized to the interventional group were given a short self-report survey at the end of each surgery (e.g. "Did the PSI go below the PSI threshold of 35 at any point during surgery?")
Postoperative delirium | Daily for three postoperative days.
  Research staff, blinded to group assignment, will assess for delirium using the Confusion Assessment Method, a physician-validated screening tool for hospital delirium

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Leung, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang CJ, Jin Z, Sands LP, Pleasants D, Tabatabai S, Hong Y, Leung JM. ADAPT-2: A Randomized Clinical Trial to Reduce Intraoperative EEG Suppression in Older Surgical Patients Undergoing Major Noncardiac Surgery. Anesth Analg. 2020 Oct;131(4):1228-1236. doi: 10.1213/ANE.0000000000004713. PMID 32925344

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT01983384/Prot_SAP_000.pdf